CLINICAL TRIAL: NCT01816724
Title: Spanish (Spain) Validation of a Specific Symptomatic Questionnaire for Patients With Nocturia
Status: Completed | Type: Observational
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, EDUARDO VICENTE PALACIO, Principal Investigator, Corporacion Parc Tauli
Other Study IDs: CSPT/URO/2013/546
Record Dates: First submitted 2013-03-20; First posted 2013-03-22 (Estimated); Last update posted 2017-06-02 (Actual); Status verified 2017-05

CONDITIONS: Nocturia
Keywords: NOCTURIA; SYMPTOMATIC QUESTIONNAIRE; N-QOL
MeSH Terms: conditions — Nocturia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Men with nocturia: Men older than 60 years old suffering from nocturia (one or more voidings overnight) without exclusion criteria
- Women with nocturia: Women older than 60 years old suffering from nocturia (one or more voidings overnight) without exclusion criteria

SUMMARY:
The objective of this study is to validate the spanish (from Spain) version of the "Nocturia Quality of Life Questionnaire and assess their psychometric properties, using the spanish translation provided by the copyright holder.

Internal consistency (measured by Alpha cronbach coefficient), Reproductibility (measured by Intraclass Correlation Coefficient), Convergent Validity (assessed using other already validate questionnaires such the International Prostate Symptom Score (IPSS), King's Health and Pittsburgh Sleeps Quality Index questionnaires) and Discriminant Validity will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Older than 60 years old
* One or more voidings overnight

Exclusion Criteria:

* Sleep disturbances
* Psychiatric diseases
* Surgical procedures during the time of study
* Introduction of new pharmacological treatments during the time of study
* Inability to complete the questionnaires

Ages: 60 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men older than 60 years old suffering from nocturia (one or more voidings overnight) without exclusion criteria
Sampling Method: Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2013-03; Primary Completion 2014-02 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
score in n-QoL questionnaire | two determinations in ten days

SECONDARY OUTCOMES:
score in IPSS spanish validated questionnaire | two determinations in ten days (only men)
score in Pittsburgh Sleep Quality Index spanish validated questionnaire | two determinations in ten days
score in King's health spanish validated questionnaire | two determinations in ten days

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Parc Tauli, Sabadell, Barcelona, Spain